CLINICAL TRIAL: NCT04958720
Title: AGAMENON-SEOM Study: Spanish Registry of Esophagogastric Cancer
Brief Title: Spanish Registry of Esophagogastric Cancer
Acronym: AGAMENON
Status: Recruiting | Type: Observational
Sponsor: Fundación Sociedad Española de Oncologia Médica (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01; RXSCXJ3E6E (Other: AEMPS)
Record Dates: First submitted 2021-06-14; First posted 2021-07-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Gastric Cancer; Gastroesophageal junction cancer; Esophageal Cancer; Surgery; Chemotherapy; Radiotherapy; Antitargeted drug; Inmunotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy; Immunotherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Resectable non-advanced cancer
  Interventions: Procedure: Surgery; Drug: Chemotherapy, anti-targeted agents and immunotherapy; Radiation: Radiotherapy
- Cohort 2: Unresectable advanced cancer
  Interventions: Procedure: Surgery; Drug: Chemotherapy, anti-targeted agents and immunotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Surgery — Surgery
Drug: Chemotherapy, anti-targeted agents and immunotherapy — Chemotherapy, anti-targeted agents and immunotherapy
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
This study aims to development of a database through a web page for epidemiological and clinical research purposes that is accessible to members of the AGAMENON - SEOM group that guarantees a rigorous collection, exploitation and analysis of the data and information contained, increases the knowledge of esophageal and stomach cancer in order to optimize the management, treatment and evolution of patients, the possibility of comparing variables with those of other series or groups, and promotes the quality of scientific publications.

DETAILED DESCRIPTION:
Patient data will be collected from medical records retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) diagnosed with carcinoma of the esophagus, gastroesophageal junction and stomach, including all histologic subtypes, with or without erbB2 overexpression (and tumors in which this data is unknown).
* Follow-up of at least 3 months with clinical information during this period, exempting patients with early death from any cause.

Exclusion Criteria:

* A patient for whom, for whatever reason, the information necessary to complete the database cannot be known or obtained.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll patients with histologically confirmed carcinoma of the esophagus, gastroesophageal junction, and stomach. The inclusion of patients is required to be done consecutively, being valid any time point if data are available.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2034-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and therapeutic approach | Up to 12 months
  To evaluate survival (time in months) according to treatment of esophagogastric cancer in all stages, patients, and contexts.

SECONDARY OUTCOMES:
Epidemiological profiles | Up to 12 months
  To know the epidemiological profiles of esophagogastric cancer in Spain: temporal and regional trends, morbidity, and mortality.
Risk factors | Up to 12 months
  To study risk factors associated with each subtype of esophagogastric cancer and localization.
Pathological features | Up to 12 months
  To evaluate the pathological features (TNM, grade, histological response)
  The TNM is measured with the American Joint Committee on Cancer (AJCC) staging system.
  The grade is classified with the WHO scale. Histological response is measured with Becker classification.
Clinical and diagnostic approach | Up to 12 months
  To know the diagnostic approch according to the center, type of studies performed: endoscopy, CT, echoendoscopy and/or PET/CT.
  From these studies it will be collected whether they have been carried out and where they visualise tumour. The use of scales and measurements is therefore not appropriate.
Treatments adjusted to prognostic variables | Up to 12 months
  To compare treatments adjusted to prognostic variables and baseline characteristics.
Validate and compare prognostic models | Up to 12 months
  To validate and compare the three prognostic models for advanced esophagogastric adenocarcinoma: The Royal Marsden Hospital index (Chau et al, 2004), and the models of Kim (2008) and Lee (2007), in a real sample of patients based on daily clinical practice.
Prognostic factors | Up to 12 months
  To analyze the prognostic factors in this population and build a predictive and/or prognostic model.
Create and validate a predictive model | Up to 12 months
  To create and validate a predictive model of early mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Dr Jiménez Fonseca, MD-PhD, Principal Investigator — Sociedad Española de Oncología Medica (SEOM)
Locations (38):
- Spain (38):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecillas, Santander, Cantabria
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Universitario de Jaén, Jaén, Jaén
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, La Coruña
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Central de la Defensa Gómez Ulla, Madrid, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Hospital Universitario de Navarra, Pamplona, Pamplona
  - Hospital Provincial de Pontevedra, Pontevedra, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario de Galdakao, Galdakao, Vizcaya

IPD SHARING:
Plan to Share IPD: No